CLINICAL TRIAL: NCT05879211
Title: Palliative Care Learning Laboratory
Brief Title: Goal Concordant Care Learning Laboratory
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00106230
Record Dates: First submitted 2023-05-14; First posted 2023-05-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Heart Failure; Copd; Dementia
Keywords: palliative care
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive; Dementia

STUDY DESIGN:
Intervention Model Description: Several interventions will be tested, at the patient and provider levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care
- Intervention (Experimental): Feedback to provider regarding frequency and quality of communication
  Interventions: Behavioral: Feedback

INTERVENTIONS:
Behavioral: Feedback — Providers will receive detailed feedback about the timing, quality, and frequency of their goals of care communication with patients
  Arms: Intervention

SUMMARY:
The goal-concordant care lab will develop and test strategies to optimize communication in advanced serious illness.

DETAILED DESCRIPTION:
The goal-concordant care lab will develop and test strategies to optimize communication in advanced serious illness. The lab will test a variety of interventions, including triggered conversations and feedback to healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Duke Health patient

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of goals of care communication | 2 years
  Frequency of goals of care conversations in the last 6 months of life
Timing of goals of care communication | 6 months
  Proximity of goals of care communication to death

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No